CLINICAL TRIAL: NCT06132100
Title: Using Wireless Transformation of Portable Three-ball Incentive Spirometers to Assist the Record of Postoperative Rehabilitation and Pulmonary Function Change in Patients Undergoing Abdominal Surgery
Brief Title: Using Digitalized Incentive Spirometers to Assist Postoperative Rehabilitation of Abdominal Surgery Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University Shuang Ho Hospital (Other)
Responsible Party: Principal Investigator, ShihChiang Shen, Visiting staff, Taipei Medical University Shuang Ho Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: N202303047
Record Dates: First submitted 2023-10-31; First posted 2023-11-15 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Bariatric Surgery Candidate; Sleep Apnea, Obstructive
Keywords: bariatric surgery; incentive spirometry
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Intervention Model Description: The purpose of this clinical trial is to use a digital recording device integrated with an incentive spirometer to record a patient's deep breathing lung training following abdominal surgery. Through this digital recording, it will be possible to effectively assess the daily frequency, duration, depth of deep breaths, and the volume of inhalation performed by the patient during their breathing exercises. This will transform the previously difficult-to-describe deep breathing training into a digital record, allowing healthcare professionals to quickly evaluate the patient's condition. Patients can also monitor their own respiratory function changes, leading to positive health promotion benefits, accelerating their postoperative recovery, and simultaneously reducing healthcare costs and improving medical quality.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigator and outcomes assessor did not know the allocation of participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- traditional incentive spirometry (Placebo Comparator): patients with traditional incentive spirometry
  Interventions: Device: traditional incentive spirometry
- digitalized incentive spirometry (Experimental): patients with digitalized incentive spirometry
  Interventions: Device: digitalized incentive spirometry

INTERVENTIONS:
Device: digitalized incentive spirometry — digitalized incentive spirometry
  Arms: digitalized incentive spirometry
Device: traditional incentive spirometry — traditional incentive spirometry
  Arms: traditional incentive spirometry

SUMMARY:
The purpose of this clinical trial is to use a digital recording device integrated with an incentive spirometer to record a patient's deep breathing lung training following abdominal surgery. Through this digital recording, it will be possible to effectively assess the daily frequency, duration, depth of deep breaths, and the volume of inhalation performed by the patient during their breathing exercises. This will transform the previously difficult-to-describe deep breathing training into a digital record, allowing healthcare professionals to quickly evaluate the patient's condition. Patients can also monitor their own respiratory function changes, leading to positive health promotion benefits, accelerating their postoperative recovery, and simultaneously reducing healthcare costs and improving medical quality.

DETAILED DESCRIPTION:
After thoracoabdominal and neurosurgery procedures, an incentive spirometer is commonly employed for deep breathing exercises to prevent or improve potential postoperative pulmonary atelectasis, increase lung capacity, promote the clearance of respiratory secretions, and maintain chest mobility to reduce postoperative complications related to lung collapse. This medical device and the respiratory training process are essential components of Enhanced Recovery After Surgery (ERAS) protocols, which integrate postoperative care processes to enhance recovery, reduce hospitalization times, and minimize postoperative complications. Currently, clinical guidelines typically recommend patients to perform 200-600 deep inhalations per day after surgery. Despite the simplicity and effectiveness of using an incentive spirometer for deep breathing exercises, the observation of patients' usage, recording of the number and duration of exercises, and tracking of their deep inhalation volumes have become crucial tasks for respiratory therapists, nurses, and physicians in the postoperative setting, consuming significant time and resources.

Generally, using an incentive spirometer requires patients to perform 200-600 deep breaths a day. According to a 2018 medical literature estimate in the United States, approximately 9.7 million surgical procedures annually involve the use of incentive spirometers, with human resource costs for assisting patients in their use and assessing the effectiveness of their pulmonary rehabilitation reaching approximately one billion US dollars.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients undergoing bariatric surgery
* 2. Patients could cooperate with conducting incentive spirometry before and after the operation.

Exclusion Criteria:

* 1. Patients with contra-indication for incentive spirometry.
* 2. Patients could not deeply breathe with pulmonary vital capacity less than 10mL/kg.
* 3. Patients could not cooperate with conducting incentive spirometry before and after the operation.
* 4. Other causes judged by the Principal Investigator

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Apnea/Hyponea Index | 7 - 10 days
  Post operative
Pulse oximetry change | 7 - 10 days
  Post operative

SECONDARY OUTCOMES:
Postoperative pulmonary complication | 7-10 days
  including atelectasis, pneumonia and respiratory failure

CONTACTS AND LOCATIONS:
Overall Officials: Shih-Chiang Shen, MD, Principal Investigator — Shung-Ho Hospital

IPD SHARING:
Plan to Share IPD: No